CLINICAL TRIAL: NCT01380080
Title: Reducing Early Mortality and Early Morbidity by Empiric Tuberculosis Treatment Regimens (REMEMBER)
Brief Title: REMEMBER: Reducing Early Mortality & Morbidity by Empiric Tuberculosis (TB) Treatment
Acronym: REMEMBER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5274; 1U01AI068636 (NIH)
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Rifampin; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Empiric (Experimental): Study treatment for Arm A participants is the strategy of initiating study-provided or other FDA-approved or tentatively approved antiretroviral treatment as soon as possible following randomization and within no more than 3 days following randomization plus a 4-drug anti-tuberculosis treatment (ATT) regimen (defined as rifampin/isoniazid/ethambutol/pyrazinamide) as soon as possible following randomization and within no more than 7 days following initiation of antiretroviral therapy. After 2 months (or 8 weeks), the 4-drug ATT will be followed with 4 months (or 16 weeks) of 2-drug ATT (defined as rifampin/isoniazid). All participants will be followed through week 96. Drug provision by or through the study will be through week 48 only
  Interventions: Drug: Atripla (r); Drug: Efavirenz; Drug: Truvada; Drug: Rifampin/isoniazid/pyrazinamide/ethambutol FDC; Drug: Rifampin/isoniazid FDC
- Arm B: IPT (Experimental): Study treatment for Arm B participants is the strategy of initiating study-provided or other FDA-approved or tentatively approved antiretroviral therapy as soon as possible following randomization and within no more than 3 days following randomization and of initiating anti-TB treatment (ATT) only when indicated according to local standard practice and at the discretion of the site investigator. All participants will be followed through week 96. Drug provision by or through the study will be through week 48 only. Pyridoxine is provided by the sites to all participants while they are receiving isoniazid (INH).
  Interventions: Drug: Atripla (r); Drug: Efavirenz; Drug: Truvada; Drug: Isoniazid

INTERVENTIONS:
Drug: Atripla (r) — Patients are administered one tablet of Efavirenz 600 mg/emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg (EFV/FTC/TDF, Atripla) to taken be taken orally once daily at bedtime without food.
Drug: Efavirenz — Participants will take one 600 mg tablet administered orally once daily without food.
  Other Names: EFV
Drug: Truvada — Participants will take one tablet of Emtricitabine 200mg/tenofovir disoproxil fumarate 300mg (FTC/TDF, Truvada) administered orally once daily with or without food.
Drug: Rifampin/isoniazid/pyrazinamide/ethambutol FDC — Participants will be administered Rifampin/isoniazid/pyrazinamide/ethambutol FDC tablets orally, once daily; dose by weight as determined in Table 5.1-1 of the protocol, for the first 8 weeks.
  Arms: Arm A: Empiric
Drug: Rifampin/isoniazid FDC — Participants will be administered rifampin/isoniazid FDC tablets orally, once daily; dose by weight as determined in Table 5.1-1 in the protocol, for 16 weeks following the first 8 weeks.
  Arms: Arm A: Empiric
Drug: Isoniazid — INH 300 mg orally once daily
  Arms: Arm B: IPT

SUMMARY:
People with HIV have a high chance of becoming infected with TB, especially when they live in areas where TB infection is common. It can be difficult to diagnose TB in people who need to start HIV treatment right away. Within about 6 months after starting HIV treatment, some of these people can become very sick with TB and can even die from it.

This study was being done in people who were starting HIV treatment and who lived in areas where the TB infection rate is high. The purpose of this study was to test an experimental approach to TB treatment to see if it is better than the usual approach. The experimental approach was to start TB treatment at the same time as HIV treatment, even when TB infection had not been found. The usual approach was to start TB treatment only if TB infection was found.

In this study, half of the people started TB treatment at the same time as they started their HIV treatment. The other half started TB treatment only if TB infection was found.

The study also tested how safe and effective it was to start TB treatment at about the same time as HIV treatment even when TB infection had not been found. The study collected information about diet, whether (and when) people in the study became sicker or died, how well their HIV was controlled, how they were feeling, how they were taking their medications, whether it mattered where they lived or what kind of HIV and TB care was standard, how many people were diagnosed with TB while in the study, and how the cost of the two treatment options on a national level could be compared.

DETAILED DESCRIPTION:
This was a randomized, open-label, phase IV strategy trial for participants from resource-limited settings (RLS) who presented with advanced HIV disease and no probable or confirmed tuberculosis (TB), and who were initiating antiretroviral treatment (ART).

Participants were randomized to one of two strategy arms: immediate, empiric TB treatment (Empiric arm) or local standard of care TB treatment (IPT arm).

Randomization was balanced by clinical trial unit and stratified according to CD4+ T cell count (<25 vs. ≥25 cells/mm^3) and presence of any of the following prognostic factors: reportable hospitalization within the past 30 days, BMI <18.5 kg/m^2, or anemia (hemoglobin <8 g/dl).

Participants were followed for 96 weeks. Participants attended study visits at screening, enrollment, and weeks 1, 2, 4, 8, 12, 16, 20, 24 and 48. Signs and symptoms, ART modifications, concomitant medications, and clinical events as defined by AIDS Clinical Trials Group (ACTG) Appendix 60 were collected at each visit. Blood was collected for CD4 and HIV-1 RNA at study entry, weeks 4, 24 and 48, and blood for safety laboratories (liver function, hematology, and renal function) was collected at all visits except week 1. A sputum sample was collected and stored at study entry. Phone contact was conducted at weeks 60, 72, 84 and 96 to obtain information about vital status, reportable hospitalization, TB status (including screening and follow-up), TB and HIV treatment modifications, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Willingness to start efavirenz-based ART as soon as possible and within no more than 3 days following randomization.
* CD4+ cell count <50 cells/mm^3 obtained within 45 days prior to study entry
* Aspartate aminotransferase (AST) (SGOT), alanine aminotransferase (ALT) (SGPT), and total bilirubin ≤ 2.5 X ULN within 30 days prior to study entry.
* Creatinine clearance ≥30 mL/min either measured or estimated using values obtained within 30 days prior to study entry.
* Results from a hepatitis B surface antigen test performed within 30 days prior to study entry.
* Agreement not to participate in a conception process (e.g., active attempt to become pregnant or to impregnate, donate sperm, in vitro fertilization).
* Female candidates of reproductive potential must have a negative serum or urine (15-25 mIU/mL) pregnancy test result within 7 days prior to study entry.
* Female candidates of reproductive potential who are participating in sexual activity that could lead to pregnancy must use two reliable methods of contraception while on study.
* Karnofsky performance score >/= 30 at time of study entry.
* Ability to swallow medications.
* Ability and willingness of participant or legal guardian/representative to provide informed consent.
* Intention to remain in the same general geographic region for the duration of study participation.

Exclusion Criteria:

* Presence of any confirmed or probable TB based on criteria listed in the current ACTG diagnosis appendix within 30 days prior to study entry and following completion of study-specific screening algorithm.
* Use of single-dose NVP for prevention of mother-to-child transmission (pMTCT) within 24 months prior to study entry.
* Use of prohibited medications within 30 days prior to study entry.
* Known allergy/sensitivity or any hypersensitivity to components of study-required ART or TB treatment.
* Current receipt of treatment for active TB or receipt of >14 days cumulative treatment for active TB within 96 weeks prior to study entry.
* Receipt of >30 days cumulative of INH prophylaxis within 48 weeks prior to study entry.
* Receipt at any time prior to study entry of >7 days cumulative treatment with any ARV or combination of ARVs (except for ARVs taken for any length of time during pregnancy for pMTCT, or ARVs taken for occupational exposure).
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Current Grade ≥2 neuropathy.
* History of multi-drug-resistant (MDR) TB.
* Within 12 weeks prior to entry, exposure to a household member or co-worker with known MDR TB.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 851 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mina C Hosseinipour, MD, Study Chair — University of North Carolina Lilongwe CRS; Johnstone Kumwenda, MBChB, FRCP, Study Chair — College of Med. JHU CRS
Locations (18):
- Instituto de Pesquisa Clinica Evandro Chagas (IPEC) CRS, Rio de Janeiro, Brazil
- Haiti (2):
  - Les Centres GHESKIO CRS, Port-au-Prince
  - GHESKIO Institute of Infectious Diseases and Reproductive Health (GHESKIO - IMIS) CRS, Port-au-Prince
- India (2):
  - YRG CARE Medical Ctr., VHS Chennai CRS, Rajiv Gandhi Salai Taramani, Chennai
  - BJ Medical College CRS, Pune, Maharashtra
- Kenya (2):
  - AMPATH at Moi Univ. Teaching Hosp. Eldoret CRS, Eldoret
  - Walter Reed Project - Kenya Med. Research Institute Kericho CRS, Kericho
- Malawi (2):
  - College of Med. JHU CRS (30301), Blantyre
  - University of North Carolina Lilongwe CRS (12001), Lilongwe
- Peru (2):
  - San Miguel CRS, San Miguel, Lima region
  - Barranco CRS (11301), Lima
- South Africa (4):
  - Wits HIV CRS, Johannesburg, Gauteng
  - CAPRISA eThekwini CRS, Durban, KwaZulu-Natal
  - Durban Adult HIV CRS, Durban, KwaZulu-Natal
  - Soweto ACTG CRS (12301), Johannesburg
- Joint Clinical Research Centre (JCRC) (12401), Kampala, Uganda
- Kalingalinga Clinic CRS (12801), Lusaka, Zambia
- UZ-Parirenyatwa CRS, AIDS Research Unit P.O. Box A178, Harare, Zimbabwe

REFERENCES:
- [Background] M. Hosseinipour, G. Bisson, S., et al. Empiric TB therapy does not decrease early mortality compared to Isoniazid Preventive therapy in adults with advanced HIV initiating ART: Results of ACTG A5274 (REMEMBER study). Program and abstracts of the 8th IAS Conference on HIV Pathogenesis, Treatment and prevention; July 19-22, 2015; Vancouver, Canada. Abstract A-729-0105-03495
- [Background] Johnstone Kumwenda, Amita Gupta, et al. Empiric TB therapy versus IPT in HIV-infected persons initiating ART (ACTG A5274 48 week results). Program and abstracts of the 2016 Conference on Retroviruses and Opportunistic Infections; February 22-25, 2016; Boston, Massachusetts. Abstract 16-1383
- [Background] Gregory P. Bisson, Amita Gupta, et al. Urine LAM Testing in Advanced HIV-Infected Adults in a Trial of Empiric TB Therapy. Program and abstracts of the 2016 Conference on Retroviruses and Opportunistic Infections; February 22-25, 2016; Boston, Massachusetts. Abstract 16-1650
- [Derived] Manabe YC, Andrade BB, Gupte N, Leong S, Kintali M, Matoga M, Riviere C, Samaneka W, Lama JR, Naidoo K, Zhao Y, Johnson WE, Ellner JJ, Hosseinipour MC, Bisson GP, Salgame P, Gupta A. A Parsimonious Host Inflammatory Biomarker Signature Predicts Incident Tuberculosis and Mortality in Advanced Human Immunodeficiency Virus. Clin Infect Dis. 2020 Dec 17;71(10):2645-2654. doi: 10.1093/cid/ciz1147. PMID 31761933
- [Derived] Hosseinipour MC, Bisson GP, Miyahara S, Sun X, Moses A, Riviere C, Kirui FK, Badal-Faesen S, Lagat D, Nyirenda M, Naidoo K, Hakim J, Mugyenyi P, Henostroza G, Leger PD, Lama JR, Mohapi L, Alave J, Mave V, Veloso VG, Pillay S, Kumarasamy N, Bao J, Hogg E, Jones L, Zolopa A, Kumwenda J, Gupta A; Adult AIDS Clinical Trials Group A5274 (REMEMBER) Study Team. Empirical tuberculosis therapy versus isoniazid in adult outpatients with advanced HIV initiating antiretroviral therapy (REMEMBER): a multicountry open-label randomised controlled trial. Lancet. 2016 Mar 19;387(10024):1198-209. doi: 10.1016/S0140-6736(16)00546-8. PMID 27025337
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009) — http://rsc.tech-res.com/safetyandpharmacovigilance/
- See also: Manual for Expedited Reporting of Adverse Events to DAID, Version 2.0, January 2010 — http://rsc.tech-res.com/clinical-research-sites/safety-reporting/manual

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited at AIDS Clinical Trials Units in 10 international countries. Recruitment occurred between October 31, 2011 (date of first participant was randomized) and June 9, 2014 (date of last participant was randomized).
Pre-assignment Details: 851 were randomized 1:1 to treatment strategies A and B. Results reported for 850 eligible participants; 1 was subsequently found ineligible and excluded from all analyses.
Period: Overall Study
Arm/Group | Arm A: Empiric | Arm B: IPT
Started | 424 | 426
Completed | 339 | 343
Not Completed | 85 | 83
Not completed — Death | 36 | 44
Not completed — Site is closing | 28 | 31
Not completed — Not able to get to clinic | 7 | 1
Not completed — Not willing to adhere to requirements | 6 | 2
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Lost to Follow-up | 3 | 3

BASELINE CHARACTERISTICS:
Population: Intent to treat: All eligible participants were included in the baseline characteristics.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Empiric | Arm B: IPT | Total
Number analyzed (Participants) | 424 | 426 | 850
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [30 to 42] | 35 [30 to 42] | 36 [30 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 200 | 400
  Male | 224 | 226 | 450
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Non-Hispanic | 375 | 384 | 759
  Hispanic (Regardless of Race) | 32 | 29 | 61
  Asian, Pacific Islander | 17 | 13 | 30
Region of Enrollment [Count of Participants; unit: Participants]
  Haiti | 53 | 56 | 109
  Malawi | 95 | 98 | 193
  Brazil | 9 | 6 | 15
  South Africa | 86 | 90 | 176
  Zimbabwe | 25 | 27 | 52
  Uganda | 25 | 24 | 49
  Zambia | 17 | 19 | 36
  Kenya | 77 | 75 | 152
  Peru | 20 | 19 | 39
  India | 17 | 12 | 29
HIV-1 RNA [Median (Inter-Quartile Range); unit: log10 copies/mL] | 5.4 [5.0 to 5.7] | 5.3 [4.9 to 5.7] | 5.3 [4.9 to 5.7]
CD4+ T-cell count [Median (Inter-Quartile Range); unit: cells/mm^3] | 18 [9 to 31] | 19 [9 to 33] | 18 [9 to 32]

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Probability of Death or Unknown Vital Status by Week 24
Description: The Kaplan-Meier estimate of the cumulative probability of death or unknown vital status by week 24.
  The vital status was considered unknown at week 24 if a participant prematurely discontinued from the study before week 24 and no vital status was obtained at week 48.
Time Frame: From study entry to week 24
Population: Intent to treat: All eligible participants were included in the analysis: participants were analyzed per original assigned randomized treatment
Measure: Number (95% Confidence Interval); unit: Cumulative probability per 100 persons
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Cumulative probability per 100 persons | 5.2 [3.5 to 7.8] | 5.2 [3.4 to 7.8]
Statistical Analysis 1: Comparison: Arm A: Empiric vs Arm B: IPT; Treatment comparison was made using the difference (arm B- arm A) in the Kaplan-Meier estimate for 24 week cumulative probability of death or unknown vital status with 95% confidence interval; Test type: Superiority or Other; p = 0.97, z-test; Cumulative probability difference = -0.06, 95% CI 2-sided [-3.05 to 2.94]

2. Secondary Outcome: Cumulative Probability of Death by Week 24
Description: The Kaplan-Meier estimate of cumulative probability of death by week 24
Time Frame: From study entry to week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Cumulative probability per 100 persons
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Cumulative probability per 100 persons | 4.8 [3.1 to 7.3] | 5.2 [3.4 to 7.8]

3. Secondary Outcome: Cumulative Probability of First AIDS Progression by Week 96
Description: The Kaplan-Meier estimate of the cumulative probability of first AIDS progression which was defined as the identification of a new World Health Organization (WHO) stage 3 or 4 condition
Time Frame: From study entry to week 96
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Cumulative probability per 100 persons
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Cumulative probability per 100 persons | 16.6 [13.3 to 20.6] | 11.3 [8.6 to 14.8]

4. Secondary Outcome: Cumulative Probability of Death or AIDS Progression by Week 24
Description: The Kaplan-Meier estimate of the cumulative probability of death or AIDS progression by week 24. AIDS progression was defined as new WHO stage 3 or 4 conditions occurred after study entry.
Time Frame: From study entry to week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Cumulative probability per 100 persons
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Cumulative probability per 100 persons | 17.1 [13.9 to 21.1] | 12.5 [9.7 to 16.0]

5. Secondary Outcome: Proportion of Participants With HIV-1 RNA Level <400 Copies/mL
Description: Proportion of participants with HIV-1 RNA level <400 copies/mL.
Time Frame: At weeks 0, 4, 24, and 48
Population: Intent to treat: All eligible participants were included in the analysis: participants were analyzed per original assigned randomized treatment. Missing data were assumed missing completed at random.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Proportion of participants
  Week 0: number analyzed (Participants) | 420 | 424
  Week 0 | 0 [0 to 0.02] | 0.01 [0 to 0.03]
  Week 4: number analyzed (Participants) | 377 | 371
  Week 4 | 0.46 [0.41 to 0.51] | 0.49 [0.44 to 0.55]
  Week 24: number analyzed (Participants) | 370 | 378
  Week 24 | 0.84 [0.79 to 0.87] | 0.85 [0.81 to 0.89]
  Week 48: number analyzed (Participants) | 361 | 366
  Week 48 | 0.87 [0.83 to 0.90] | 0.89 [0.86 to 0.92]

6. Secondary Outcome: CD4+ T-cell Count
Description: The absolute levels of CD4+ T-cell counts (cells/mm^3)
Time Frame: At weeks 0, 4, 24, and 48
Population: Intent to treat: All eligible participants were included in the analysis: Participants were analyzed per original assigned randomized treatment. Missing data were assigned missing completely at random.
Measure: Median (Inter-Quartile Range); unit: cells/ mm^3
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
cells/ mm^3
  Week 0: number analyzed (Participants) | 422 | 425
  Week 0 | 18 [9 to 31] | 19 [9 to 33]
  Week 4: number analyzed (Participants) | 406 | 406
  Week 4 | 74 [37 to 118] | 76 [41 to 123]
  Week 24: number analyzed (Participants) | 387 | 393
  Week 24 | 121 [75 to 172] | 121 [80 to 188]
  Week 48: number analyzed (Participants) | 362 | 364
  Week 48 | 176 [112 to 251] | 172 [112 to 245]

7. Secondary Outcome: CD4+ T-cell Count Change From Baseline
Description: Change was calculated as the CD4+ T-cell count at the later weeks (4, 24 and 48) minus the baseline (week 0) CD4+ T-cell count.
Time Frame: Weeks 0, 4, 24 and 48
Population: Intention to treat: All eligible participants were included in the analysis: participants were analyzed per original assigned randomized treatment. Missing data were assumed missing completely at random.
Measure: Median (Inter-Quartile Range); unit: cells/ mm^3
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
cells/ mm^3
  Week 4: number analyzed (Participants) | 404 | 405
  Week 4 | 49 [20 to 91] | 54 [22 to 94]
  Week 24: number analyzed (Participants) | 385 | 392
  Week 24 | 96 [55 to 147] | 102 [60 to 159]
  Week 48: number analyzed (Participants) | 360 | 364
  Week 48 | 158 [92 to 224] | 146 [90 to 219]

8. Secondary Outcome: Time to Initiation of TB Treatment by Week 96
Description: Median time to TB treatment initiation since study entry
Time Frame: From study entry to week 96
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Days | 0 [0 to 1] | 0 [0 to 1]

9. Secondary Outcome: Proportion of Participants With TB Diagnosis by Week 96
Description: Proportion of participants with TB diagnosis per current ACTG Diagnosis Appendix 60 by week 96
Time Frame: From study entry to week 96
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Proportion of participants | 0.08 | 0.05

10. Secondary Outcome: Proportion of Participants With at Least One New Grade 3 or 4 Adverse Event That is at Least a One-grade Increase From Baseline by Week 48
Description: Proportion of participants with at least one new Grade 3 or 4 laboratory or sign or symptom that is at least a one-grade increase from baseline by Week 48. Grade 3=Severe, Grade 4=Life-Threatening according to DAIDS AE Grading Table (see references).
Time Frame: From study entry to week 48
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Proportion of participants | 0.32 | 0.30

11. Secondary Outcome: Proportion of Participants With at Least One New Grade 3 or 4 Targeted Laboratory Value That is at Least a One-grade Increase From Baseline by Week 48
Description: Proportion of participants with at least one new Grade 3 or 4 that is at least a one-grade increase from baseline for the following targeted laboratory values by Week 48
  The targeted laboratory events include hemoglobin, serum creatinine, ALT and AST
Time Frame: From study entry to week 48. The lab events were collected at study entry, weeks 2, 4, 8, 12, 16, 20, 24, and 48.
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Proportion of participants | 0.11 | 0.13

12. Secondary Outcome: Proportion of Participants With Immune Reconstitution Inflammatory Syndrome (IRIS) by Week 48
Description: Proportion of participants with IRIS (using current ACTG definition Appendix 60, see References) by Week 48. IRIS in participants with TB and other opportunistic infections may occur shortly after the initiation of potent combination ART, particularly in participants with advanced HIV disease.
Time Frame: From study entry to week 48
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Proportion of participants | 0.04 | 0.05

13. Secondary Outcome: Proportion of Participants With Reportable Hospitalization by Week 48
Description: Proportion of participants with reportable hospitalization reported by Week 48
Time Frame: From study entry to week 48
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Proportion of participants | 0.10 | 0.12

14. Secondary Outcome: Proportion of Participants Who Prematurely Discontinued Any Component of TB Treatment by Week 48
Description: Proportion of participants with premature discontinuation of any component of TB treatment by Week 48
Time Frame: From study entry to week 48
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Proportion of participants | 0.13 | 0.05

15. Secondary Outcome: Proportion of Participants Who Prematurely Discontinued Antiretroviral Therapy by Week 48
Description: Proportion of participants with premature discontinuation of antiretroviral therapy (ART) by Week 48
Time Frame: From study entry to week 48
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Proportion of participants | 0.19 | 0.21

16. Secondary Outcome: Cumulative Probability of Death or AIDS Progression by Week 48
Description: The Kaplan-Meier estimate of the cumulative probability of death or AIDS progression by week 48. AIDS progression was defined as new WHO stage 3 or 4 conditions occurred after study entry.
Time Frame: From study entry to week 48
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Cumulative probability per 100 persons
Arm/Group | Arm A: Empiric | Arm B: IPT
Number analyzed (Participants) | 424 | 426
Cumulative probability per 100 persons | 19.3 [15.8 to 23.4] | 15.3 [12.2 to 19.1]

ADVERSE EVENTS:
Time Frame: From treatment dispensation to up to week 96
Description: The protocol required reporting of signs and symptoms and laboratory abnormalities of >=Grade 2 and all grades of fever. The DAIDS AE Grading Table (V1.0) and EAE Manual (V2.0) were used.
Arm/Group | Arm A: Empiric | Arm B: IPT
All-Cause Mortality (participants affected / at risk) | 36/424 | 44/426
Serious Adverse Events (participants affected / at risk) | 85/424 | 94/426
Other Adverse Events (participants affected / at risk) | 380/424 | 379/426
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Empiric (N=424) | Arm B: IPT (N=426)
Anaemia (Blood and lymphatic system disorders) | 7 | 7
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Death (General disorders) | 2 | 8
Multi-organ failure (General disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 4 | 3
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Acquired immunodeficiency syndrome (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Central nervous system infection (Infections and infestations) | 0 | 1
Cerebral toxoplasmosis (Infections and infestations) | 1 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1
Disseminated tuberculosis (Infections and infestations) | 2 | 1
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 6 | 6
HIV infection (Infections and infestations) | 0 | 1
Histoplasmosis disseminated (Infections and infestations) | 1 | 0
Immune reconstitution inflammatory syndrome associated tuberculosis (Infections and infestations) | 1 | 0
Lymph node tuberculosis (Infections and infestations) | 2 | 0
Malaria (Infections and infestations) | 3 | 2
Meningitis (Infections and infestations) | 1 | 1
Meningitis bacterial (Infections and infestations) | 0 | 2
Meningitis cryptococcal (Infections and infestations) | 6 | 9
Meningitis tuberculous (Infections and infestations) | 1 | 5
Meningitis viral (Infections and infestations) | 1 | 1
Neurosyphilis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 7 | 3
Pneumonia bacterial (Infections and infestations) | 5 | 3
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Salmonella sepsis (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 2 | 4
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tuberculoma of central nervous system (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 4 | 1
Typhoid fever (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Viral vasculitis (Infections and infestations) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 3 | 1
Weight decreased (Investigations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 2
Hallucination (Psychiatric disorders) | 1 | 0
Reactive psychosis (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Abortion induced (Surgical and medical procedures) | 1 | 0
Cryptococcal fungaemia (Infections and infestations) | 1 | 0
HIV-associated neurocognitive disorder (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Empiric (N=424) | Arm B: IPT (N=426)
Abdominal pain (Gastrointestinal disorders) | 28 | 26
Diarrhoea (Gastrointestinal disorders) | 42 | 34
Nausea (Gastrointestinal disorders) | 22 | 22
Vomiting (Gastrointestinal disorders) | 39 | 51
Pyrexia (General disorders) | 46 | 55
Oral candidiasis (Infections and infestations) | 49 | 49
Pulmonary tuberculosis (Infections and infestations) | 22 | 13
Alanine aminotransferase increased (Investigations) | 58 | 75
Aspartate aminotransferase increased (Investigations) | 99 | 101
Blood albumin decreased (Investigations) | 151 | 159
Blood alkaline phosphatase increased (Investigations) | 36 | 43
Blood bicarbonate decreased (Investigations) | 66 | 72
Blood creatinine increased (Investigations) | 25 | 45
Blood potassium decreased (Investigations) | 32 | 31
Blood sodium decreased (Investigations) | 144 | 140
Haemoglobin decreased (Investigations) | 119 | 95
Neutrophil count decreased (Investigations) | 161 | 163
Platelet count decreased (Investigations) | 32 | 38
Weight decreased (Investigations) | 34 | 25
White blood cell count decreased (Investigations) | 136 | 130
Headache (Nervous system disorders) | 27 | 43
Vaginal discharge (Reproductive system and breast disorders) | 22 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 48
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 43 | 32
Anaemia (Blood and lymphatic system disorders) | 21 | 22
Chest pain (General disorders) | 18 | 22
Pneumonia bacterial (Infections and infestations) | 23 | 21
Blood sodium increased (Investigations) | 22 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 23
Rash (Skin and subcutaneous tissue disorders) | 21 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.